CLINICAL TRIAL: NCT00312377
Title: A Phase III, Randomized, Double-Blinded, Multi-Center, Study to Assess the Efficacy of Docetaxel (TAXOTERE™) in Combination With ZD6474 (ZACTIMA™) Versus Docetaxel (TAXOTERE™) With Placebo in Subjects With Locally Advanced or Metastatic NSCLC
Brief Title: ZACTIMA (an Anti-EGFR / Anti-VEGF Agent) Combined With Docetaxel Compared to Docetaxel in Non-small Cell Lung Cancer
Acronym: ZODIAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00032; 6474IL/0032; 2005-004749-32 (EudraCT Number)
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer
Keywords: Non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel; vandetanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Docetaxel monotherapy
  Interventions: Drug: Docetaxel
- 2 (Experimental): Vandetanib + Docetaxel
  Interventions: Drug: Docetaxel; Drug: Vandetanib

INTERVENTIONS:
Drug: Docetaxel — infusion
  Other Names: TAXOTERE™
Drug: Vandetanib — oral
  Other Names: ZACTIMA™; ZD6474
  Arms: 2

SUMMARY:
This large phase III clinical study is studying the effect of vandetanib (ZACTIMA) in treating non-small cell lung cancer (NSCLC). Vandetanib is a new type of agent that targets the blood supply to a cancer tumour (through it's anti-vascular endothelial growth factor receptor (VEGFR) properties) and the tumour cells themselves (through it's anti-endothelial growth factor receptor (EGFR) actions). This study will look at the effects of vandetanib in lung cancer patients who have had their cancer re-appear after treatment with standard chemotherapy.

This clinical study will test if the vandetanib anti-VEGF and anti-EGFR characteristics can deliver longer improved progression free survival and improved overall survival than docetaxel (Taxotere) alone.

All patients participating this clinical study will receive treatment with docetaxel, a commonly used treatment for recurrent non-small cell lung cancer.

In addition, some patients will also receive vandetanib (ZACTIMA), an anti-EGFR / anti-VEGF agent.

Recent clinical research shows that vascular endothelial growth factor receptor (VEGFR) inhibition, when used with standard chemotherapy, can lead to increased survival in advanced non-small cell lung cancer (NSCLC) patients.

Other research shows that epidermal growth factor receptor (EGFR) inhibitors, like erlotinib (Tarceva) can also increase overall non-small cell lung cancer survival by killing tumour cells and stopping them from dividing.

ELIGIBILITY:
Inclusion Criteria:

Lung cancer patients who answer true to the following statements are eligible to join this clinical study.

* I have a confirmed diagnosis of locally advanced or metastatic non small cell lung cancer (Stage IIIb - IV)
* I have had 1st line anti-cancer therapy. Previous treatment with Avastin (bevacizumab) in first line NSCLC is allowed.

Exclusion Criteria:

Lung cancer patients who answer true to the following are NOT eligible to join this clinical study.

* I do not have non small cell lung cancer (NSCLC)
* I have received treatment with docetaxel (Taxotere). Prior treatment with paclitaxel is acceptable.
* I have received 2nd line anti-cancer therapy (For example, patients with previous 2nd line non small cell lung cancer (NSCLC) treatment with Tarceva (erlotinib, OSI-744), Alimta (pemetrexed) are not eligible)
* I have been treated with VEGFR-tyrosine kinase inhibitors (TKIs) (sunitinib, sorafenib, other VEGF TKIs). Previous treatment with Avastin (bevacizumab) in 1st line non small cell lung cancer is permitted.
* I have a history of uncontrolled irregular heartbeat
* I have a history of high blood pressure which has not been controlled with medication If you are unsure of the meaning of the inclusion and exclusion criteria above, please contact the call center number for help.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1690 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Contact-US@sanofi.com, Study Director — Sanofi
Locations (156):
- United States (27):
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Norwalk, Connecticut
  - Research Site, Ocala, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Joliet, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Hutchinson, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Albany, New York
  - Research Site, Armonk, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Ogden, Utah
  - Research Site, Alexandria, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Vancouver, Washington
- Argentina (5):
  - Research Site, Bahía Blanca
  - Research Site, Capital Federal
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Mendoza
  - Research Site, Rosario
- Austria (6):
  - Research Site, Graz
  - Research Site, Grimmenstein
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (5):
  - Research Site, Brussels (Jette)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Edegem
  - Research Site, Genk
  - Research Site, Liège
- Brazil (5):
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Québec, Quebec
- China (6):
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan
- Denmark (5):
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Odense
  - Research Site, Roskilde
  - Research Site, Vejle
- France (8):
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Nancy
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Herblain
- Germany (11):
  - Research Site, Bad Berka
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Oldenburg
  - Research Site, Ulm
  - Research Site, Wiesbaden
- Greece (2):
  - Research Site, Athens
  - Research Site, Heraklion
- India (7):
  - Research Site, Ahmedabad
  - Research Site, Chennai
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vellore
- Indonesia (2):
  - Research Site, Jakarta Timur
  - Research Site, Yogyakarta
- Italy (11):
  - Research Site, Ancona
  - Research Site, Avellino
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Mantova
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Reggio Emilia
- Japan (20):
  - Research Site, Akashi-shi
  - Research Site, Fukuoka
  - Research Site, Isehara-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Okazaki-shi
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Toyonaka
  - Research Site, Ube-shi
  - Research Site, Utsunomiya
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, George Town
  - Research Site, Kampung Baharu Nilai
  - Research Site, Kubang Kerian
- Mexico (3):
  - Research Site, Durango
  - Research Site, Morelia
  - Research Site, Toluca
- Netherlands (4):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Maastricht
- Portugal (5):
  - Research Site, Coimbra
  - Research Site, Funchal
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Research Site, Singapore, Singapore
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Zaragoza
- Research Site, Chiang Mai, Thailand
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Lombard A, Mistry H, Aarons L, Ogungbenro K. Dose individualisation in oncology using chemotherapy-induced neutropenia: Example of docetaxel in non-small cell lung cancer patients. Br J Clin Pharmacol. 2021 Apr;87(4):2053-2063. doi: 10.1111/bcp.14614. Epub 2020 Dec 19. PMID 33075149
- [Derived] Platt A, Morten J, Ji Q, Elvin P, Womack C, Su X, Donald E, Gray N, Read J, Bigley G, Blockley L, Cresswell C, Dale A, Davies A, Zhang T, Fan S, Fu H, Gladwin A, Harrod G, Stevens J, Williams V, Ye Q, Zheng L, de Boer R, Herbst RS, Lee JS, Vasselli J. A retrospective analysis of RET translocation, gene copy number gain and expression in NSCLC patients treated with vandetanib in four randomized Phase III studies. BMC Cancer. 2015 Mar 23;15:171. doi: 10.1186/s12885-015-1146-8. PMID 25881079
- [Derived] Heymach JV, Lockwood SJ, Herbst RS, Johnson BE, Ryan AJ. EGFR biomarkers predict benefit from vandetanib in combination with docetaxel in a randomized phase III study of second-line treatment of patients with advanced non-small cell lung cancer. Ann Oncol. 2014 Oct;25(10):1941-1948. doi: 10.1093/annonc/mdu269. Epub 2014 Jul 23. PMID 25057173
- [Derived] Herbst RS, Sun Y, Eberhardt WE, Germonpre P, Saijo N, Zhou C, Wang J, Li L, Kabbinavar F, Ichinose Y, Qin S, Zhang L, Biesma B, Heymach JV, Langmuir P, Kennedy SJ, Tada H, Johnson BE. Vandetanib plus docetaxel versus docetaxel as second-line treatment for patients with advanced non-small-cell lung cancer (ZODIAC): a double-blind, randomised, phase 3 trial. Lancet Oncol. 2010 Jul;11(7):619-26. doi: 10.1016/S1470-2045(10)70132-7. PMID 20570559
- See also: CSR-D4200C00032.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=340&filename=CSR-D4200C00032.pdf
- See also: CSP Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=340&filename=vandetanib_Study_32_ZODIAC_CSP_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 08 May 2006, last patient enrolled 14 March 2008, cut off date 22 August 2008
Groups:
- Vandetanib 100 mg Plus Docetaxel: Vandetanib 100 mg oral tablet taken once daily in combination with docetaxel 75 mg/m2 IVb infusion every 21 days up to a maximum of 6 cycles
- Placebo Plus Docetaxel: Placebo tablet taken once daily plus docetaxel 75 mg/m2 IVb infusion every 21 days up to a maximum of 6 cycles
Period: Overall Study
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Started | 694 (randomised patients) | 697 (randomised patients)
Completed | 50 (ongoing study treatment at data cut-off) | 29 (ongoing study treatment at data cut-off)
Not Completed | 644 | 668
Not completed — Death | 403 | 418
Not completed — Withdrawal by Subject | 23 | 30
Not completed — Lost to Follow-up | 9 | 12
Not completed — Non-compliance | 0 | 2
Not completed — Randomised but never received treatment | 6 | 6
Not completed — Discontinue treatment survival follow up | 202 | 200
Not completed — Site ended participation in study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vandetanib 100 mg Plus Docetaxel: Vandetanib 100 mg plus docetaxel
- Placebo Plus Docetaxel: Placebo plus docetaxel
- Total: Total of all reporting groups
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel | Total
Number analyzed (Participants) | 694 | 697 | 1391
Age, Continuous [Mean (Full Range); unit: years] | 58.5 [28 to 82] | 58.4 [20 to 82] | 58.45 [20 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 497 | 473 | 970
  Male | 197 | 224 | 421

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) in the Overall Population
Description: Median time (in weeks) from randomisation until objective disease progression or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable RECIST assessment. Progression was derived according to RECIST 1.0 and is defined as an increase of at least 20% in the total tumour size of measurable lesions over the nadir measurement, unequivocal progression in the non-target lesions or the appearance of one or more new lesions.
Time Frame: RECIST tumour assessments carried out every 6 weeks from randomisation until the date of first documented objective disease progression or date of death from any cause, whichever came first assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 694 | 697
Weeks | 17.3 [15 to 18] | 14 [12.7 to 16.9]

2. Primary Outcome: Progression-Free Survival (PFS) in the Female Population
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 197 | 224
Weeks | 20.1 [17.9 to 23.9] | 18.3 [15 to 22.1]

3. Secondary Outcome: Overall Survival (OS) in the Overall Population
Description: Overall survival is defined as the time from date of randomization until death. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive (ie their status must be known at the censored date and should not be lost to follow up or unknown).
Time Frame: Time to death in months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 694 | 697
Months | 10.6 [9.6 to 11.5] | 10 [9.2 to 10.8]

4. Secondary Outcome: Overall Survival (OS) in the Female Population
Description: as for outcome 3
Time Frame: Time to death in months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 197 | 224
Months | 12.7 [10.5 to 17.1] | 14.2 [10.8 to 16.2]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the number of patients that are responders ie those patients with a confirmed best objective response of complete response (CR) or partial response (PR) as determined according to RECIST 1.0. CR is defined as the disappearance of all target lesions with no evidence of tumour elsewhere and PR is defined as at least a 30% reduction in the total tumour size of measurable lesions with no new lesions and no progression in the non-target lesions.
Time Frame: Each patient was assessed for objective response from the sequence of RECIST scan data up to data cut off. RECIST tumour assessments carried out every 6 weeks from randomisation until objective progression
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 694 | 697
Participants | 120 | 71

6. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is defined as the number of patients who achieved disease control at least 6 weeks following randomisation. Disease control at 6 weeks is defined as a best objective response of complete response (CR), partial response (PR) or stable disease (SD) >= 6 weeks as determined according to RECIST 1.0. CR is defined as the disappearance of all target lesions with no evidence of tumour elsewhere, PR is defined as at least a 30% reduction in the total tumour size of measurable lesions with no new lesions and no progression in the non-target lesions and SD >= 6 is assigned to patients who have not responded and have no evidence of progression at least 6 weeks after randomisation.
Time Frame: RECIST tumour assessments carried out every 6 weeks from randomisation until objective progression
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 694 | 697
Participants | 413 | 380

7. Secondary Outcome: Duration of Response (DoR)
Description: Response is defined as a confirmed best objective response of CR or PR. Duration of response is defined as time from the date of first documented response until date of documented progression or death in the absence of disease progression (provided death is within 3 months of last RECIST assessment)
Time Frame: RECIST tumour assessments carried out every 6 weeks from randomisation until objective progression
Measure: Median (Full Range); unit: Weeks
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 694 | 697
Weeks | 29.9 [7.14 to 72.29] | 19.7 [9.71 to 41.86]

8. Secondary Outcome: Time to Deterioration of Disease-related Symptoms (TDS) by Functional Assessment of Cancer Therapy - Lung (FACT-L) Lung Cancer Subscale (LCS).
Description: The lung cancer subscale (LCS) consists of 7 items of the FACT-L (3 items relating to breathing/dyspnea, and 1 item each relating to cough, weight loss, appetite, and cognition). The LCS total score is the sum of the scores from the 7 items.
  Time to deterioration is defined as the interval from the date of randomization to the first assessment of worsened without an improvement in the next 21 days.
  A patient will be defined as having a deterioration in symptoms if they have a single visit assessment of 'worsened' with no visit assessment of 'improved' within the next 21 days.
Time Frame: FACT-L questionnaires are to be administered every 3 weeks after randomisation
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 694 | 697
Weeks | 15 [6.1 to 82.3] | 11.9 [6.0 to 28.1]

9. Secondary Outcome: Time to Deterioration of Disease-related Symptoms (TDS) by FACT-L Pulmonary Symptom Index (PSI)
Description: The pulmonary symptom index (PSI) consists of 4 items of the LCS relating to pulmonary symptoms (i.e. 3 items relating to breathing/dyspnea, and 1 item relating to cough). The PSI score is the sum of the scores from the 4 items.
  Time to deterioration is defined as the interval from the date of randomization to the first assessment of worsened without an improvement in the next 21 days.
  A patient will be defined as having a deterioration in symptoms if they have a single visit assessment of 'worsened' with no visit assessment of 'improved' within the next 21 days.
Time Frame: FACT-L questionnaires are to be administered every 3 weeks after randomisation
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 694 | 697
Weeks | 12.3 [5.9 to 36.7] | 11.9 [6 to 28.4]

ADVERSE EVENTS:
Arm/Group | Vandetanib 100 mg Plus Docetaxel | Placebo Plus Docetaxel
Serious Adverse Events (participants affected / at risk) | 263/694 | 232/697
Other Adverse Events (participants affected / at risk) | 637/694 | 630/697
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg Plus Docetaxel (N=694) | Placebo Plus Docetaxel (N=697)
Febrile Neutropenia (Blood and lymphatic system disorders) | 46 | 38
Neutropenia (Blood and lymphatic system disorders) | 16 | 18
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 3 | 10
Myocardial Infarction (Cardiac disorders) | 0 | 4
Cardiac Arrest (Cardiac disorders) | 1 | 3
Cardiac Failure (Cardiac disorders) | 0 | 3
Acute Myocardial Infarction (Cardiac disorders) | 2 | 2
Atrial Flutter (Cardiac disorders) | 2 | 1
Angina Unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1
Hereditary Angioedema (Congenital, familial and genetic disorders) | 1 | 0
Deafness Unilateral (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ocular Surface Disease (Eye disorders) | 1 | 0
Retinal Artery Occlusion (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 11
Vomiting (Gastrointestinal disorders) | 7 | 8
Nausea (Gastrointestinal disorders) | 5 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Gastric Ulcer (Gastrointestinal disorders) | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0
Appendicitis Perforated (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal Fistula (Gastrointestinal disorders) | 1 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 1 | 0
Proctitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 13 | 12
Asthenia (General disorders) | 2 | 5
Chest Pain (General disorders) | 3 | 0
Malaise (General disorders) | 3 | 0
Performance Status Decreased (General disorders) | 3 | 0
Fatigue (General disorders) | 1 | 2
General Physical Health Deterioration (General disorders) | 1 | 2
Mucosal Inflammation (General disorders) | 1 | 2
Chills (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 1
Anaphylactic Shock (Immune system disorders) | 1 | 2
Drug Hypersensitivity (Immune system disorders) | 2 | 1
Pneumonia (Infections and infestations) | 33 | 26
Respiratory Tract Infection (Infections and infestations) | 5 | 6
Sepsis (Infections and infestations) | 5 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 5
Gastroenteritis (Infections and infestations) | 4 | 3
Lung Infection (Infections and infestations) | 4 | 2
Urinary Tract Infection (Infections and infestations) | 4 | 3
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 1
Septic Shock (Infections and infestations) | 3 | 1
Bacterial Infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 0 | 2
Neutropenic Infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial Sepsis (Infections and infestations) | 1 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 | 0
Catheter Related Infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Central Line Infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 1
Infective Myositis (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Lung Abscess (Infections and infestations) | 1 | 1
Oesophageal Candidiasis (Infections and infestations) | 1 | 0
Perianal Abscess (Infections and infestations) | 0 | 1
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 1 | 0
Rash Pustular (Infections and infestations) | 1 | 0
Rectal Abscess (Infections and infestations) | 1 | 0
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Skin Bacterial Infection (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 2
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 1
Weight Decreased (Injury, poisoning and procedural complications) | 0 | 2
White Blood Cell Count Decreased (Injury, poisoning and procedural complications) | 0 | 2
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 0 | 1
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 0 | 1
Blood Alkaline Phosphatase Increased (Injury, poisoning and procedural complications) | 0 | 1
Blood Pressure Orthostatic Decreased (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram T Wave Abnormal (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 1 | 3
Loss Of Consciousness (Nervous system disorders) | 3 | 1
Somnolence (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 2 | 2
Altered State Of Consciousness (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Brachial Plexopathy (Nervous system disorders) | 0 | 1
Cauda Equina Syndrome (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Coma Hepatic (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Pyramidal Tract Syndrome (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Psychotic Behaviour (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2
Renal Failure (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 21
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cryptogenic Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic Rupture (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 15 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 5 | 0
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 4 | 0
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 3 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 3 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 2 | 0
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 6
Hypotension (Vascular disorders) | 5 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0
Superior Vena Caval Stenosis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Vena Cava Thrombosis (Vascular disorders) | 0 | 1
Venous Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg Plus Docetaxel (N=694) | Placebo Plus Docetaxel (N=697)
Neutropenia (Blood and lymphatic system disorders) | 212 | 174
Leukopenia (Blood and lymphatic system disorders) | 125 | 106
Anaemia (Blood and lymphatic system disorders) | 68 | 98
Diarrhoea (Gastrointestinal disorders) | 284 | 218
Nausea (Gastrointestinal disorders) | 158 | 221
Vomiting (Gastrointestinal disorders) | 105 | 141
Constipation (Gastrointestinal disorders) | 119 | 140
Stomatitis (Gastrointestinal disorders) | 80 | 80
Abdominal Pain (Gastrointestinal disorders) | 41 | 50
Dyspepsia (Gastrointestinal disorders) | 37 | 25
Abdominal Pain Upper (Gastrointestinal disorders) | 30 | 36
Fatigue (General disorders) | 208 | 214
Pyrexia (General disorders) | 127 | 110
Asthenia (General disorders) | 105 | 90
Oedema Peripheral (General disorders) | 49 | 57
Mucosal Inflammation (General disorders) | 49 | 38
Nasopharyngitis (Infections and infestations) | 41 | 37
Weight Decreased (Infections and infestations) | 54 | 41
Anorexia (Metabolism and nutrition disorders) | 199 | 204
Myalgia (Musculoskeletal and connective tissue disorders) | 90 | 78
Back Pain (Musculoskeletal and connective tissue disorders) | 51 | 62
Arthralgia (Musculoskeletal and connective tissue disorders) | 61 | 52
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 39 | 31
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 35 | 30
Headache (Nervous system disorders) | 58 | 62
Dizziness (Nervous system disorders) | 43 | 58
Dysgeusia (Nervous system disorders) | 40 | 49
Peripheral Sensory Neuropathy (Nervous system disorders) | 42 | 48
Paraesthesia (Nervous system disorders) | 42 | 42
Insomnia (Psychiatric disorders) | 95 | 73
Cough (Respiratory, thoracic and mediastinal disorders) | 130 | 133
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 102 | 122
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 50 | 27
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 37 | 45
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 41 | 20
Hiccups (Respiratory, thoracic and mediastinal disorders) | 30 | 41
Rash (Skin and subcutaneous tissue disorders) | 282 | 166
Alopecia (Skin and subcutaneous tissue disorders) | 230 | 240
Pruritus (Skin and subcutaneous tissue disorders) | 65 | 42
Nail Disorder (Skin and subcutaneous tissue disorders) | 52 | 46
Dry Skin (Skin and subcutaneous tissue disorders) | 45 | 30
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 42 | 1
Hypertension (Vascular disorders) | 41 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.